CLINICAL TRIAL: NCT05346198
Title: A Phase I Clinical Trial to Evaluate CART-BCMA in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Evaluate CART-BCMA in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B03B00301-101
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects will receive CART-BCMA (Experimental): Biological: CART-BCMA Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to produce CART-BCMA.
  During CART-BCMA production, subjects may receive bridging chemotherapy for disease control. Upon successful generation of CART-BCMA product, subjects will receive treatment with CART-BCMA therapy.
  Study treatment will include lymphodepleting chemotherapy followed by one dose of CART-BCMA administered by intravenous (IV) injection.
  Interventions: Drug: CART-BCMA

INTERVENTIONS:
Drug: CART-BCMA — The CART-BCMA (study drug) used in this study are chimeric antigen receptor specifically expressing T cells targeting BCMA.

SUMMARY:
This is a Phase 1, multicenter, open-label study o evaluate the safety and efficacy of CART-BCMA in subjects with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
The study will consist of 2 parts: dose-escalation (Part A) and dose-expansion (Part B). The dose-escalation part (Part A) of the study is to evaluate the safety and tolerability of increasing dose levels of CART-BCMA to establish a recommended dose (RD); and the dose-expansion part (Part B) of the study is to further evaluate the safety, pharmacokinetics/pharmacodynamics, and efficacy of CART-BCMA at the RD.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old (inclusive), gender is not limited;
* Multiple myeloma patients who have received at least 3-line previous multiple myeloma therapy and have failed at least through proteasome inhibitors and immunomodulators; Each line of treatment has at least 1 complete treatment cycle, unless the best remission for the treatment is recorded as disease progression (PD) (according to the IMWG Efficacy Evaluation Criterialpublished in 2016, Appendix 4); PD must be recorded during or within 12 months after the last treatment;
* Bone marrow specimens were confirmed by immunohistochemistry or flow cytometry as positive BCMA expression in plasma cells and myeloma cells (>5%);
* The presence of measurable lesions during screening was defined as any of the following:

Serum M protein ≥1 g/dL (≥10 g/L); Urinary M protein level ≥200 mg/24 h; Serum light chain (FLC) : abnormal serum FLC ratio (< 0.26 or > 1.65), and affected FLC≥10 mg/dL (100mg/L);

* ECOG score (Appendix 1) 0~1;
* Expected survival time ≥3 months;
* The mononuclear cells meet the following standards within 3 days before collection:

Hematology:≥0.5×109/L[The use of past granulocyte colony stimulating factor (G-CSF) is allowed, but patients shall not receive this supportive treatment within 7 days prior to the screening phase of laboratory examination];≥1.0 ×109 /L[Ex-granulocyte colony-stimulating factor (G-CSF) is allowed, but subjects shall not receive this supportive treatment within 7 days prior to the screening laboratory examination];Subjects' platelet count ≥50×109/L (Subjects shall not receive blood transfusion support within 7 days before the screening laboratory examination);≥8.0 g/dL (Recombinant Human Erythropoietin is allowed) [Subjects have not received a red blood cell infusion (RBC) within 7 days prior to the screening phase laboratory examination]; Heart:Left ventricular ejection fraction (LVEF) ≥ 50%; Lung:Blood oxygen saturation ≥91% under non-inhaled oxygen condition; Kidney:Creatinine clearance (CRCL) or glomerular filtration rate (GFR) (Cockcroft-Gault formula) ≥30 mL/min; Liver:Total bilirubin (serum) ≤1.5 × ULN;Gilbert's disease patients with >1.5 × ULN could be enrolled with the consent of the Sponsor; Blood coagulation:Plasma prothrombin time (PT) ≤1.5 × ULN, international standardized ratio (INR) ≤1.5 × ULN, partial prothrombin time (APTT) ≤1.5 × ULN;

* Peripheral venous access can meet the needs of single collection and intravenous drip;
* The subject agrees to use reliable contraceptive methods for contraception within 1 year after signing the informed consent form to the infusion. Including but not limited to: abstinence, men undergoing vasectomy, implantable progesterone contraceptives that can inhibit ovulation; intrauterine contraceptive devices; hormone-releasing intrauterine devices; sexual partner sterilization methods; copper intrauterine devices, Correct use of proven compound hormonal contraceptives that can inhibit ovulation; progesterone contraceptives that can inhibit ovulation. At the same time, female subjects should promise not to donate eggs (egg cells, oocytes) for assisted reproduction within 1 year after the infusion;
* Volunteer to participate in clinical trials and sign Informed Consent Form;

Exclusion Criteria:

* Subjects who are known to have allergic reactions, hypersensitivity, intolerance, or contraindications to any component of CART-BCMA or any drugs that may be used in the study (including fludarabine, cyclophosphaamide, or tozumab), or who are allergic to β-lactam antibiotics, or who have had severe allergic reactions in the past;
* Prior to any CAR-T therapy or BCMA-targeted therapy;
* Have received the following anti-MM treatment within the prescribed time range before single calyzer:

Has received small molecule targeted therapy within 4 weeks or 5 half-lives, whichever is longer; treatment with a large molecule within 4 weeks or 2 half-lives, whichever is longer; received cytotoxic therapy, proteasome inhibitor, or modern Chinese medicine preparation with anti-tumor effect within 2 weeks; received immunomodulatory drug therapy within 1 week; received radiotherapy within 1 week

* Participated in a clinical trial within 4 weeks before the single collection;
* Patients who received autologous hematopoietic stem cell transplantation (ASCT) or previous allogeneic stem cell transplantation within 12 weeks before a single collection (no time limit);
* People who received live vaccine or attenuated vaccine within 4 weeks before the CART-BCMA harvest; Note: Inactivated viral vaccines for seasonal influenza are allowed for injection; Intranasally administered live attenuated influenza vaccines are not allowed;
* Received any of the following treatments within 7 days prior to the single collection or as determined by the investigator to require long-term treatment during the study period:

Systemic steroid therapy (except inhalation or topical use), Immunosuppressive therapy, Graft versus host therapy, Preventive treatment of central nervous system

* Incomplete recovery or stabilization to grade 1 (NCI-CTCAE v5.0) of toxicity (including peripheral neuropathy) caused by previous treatment;
* MM is suspected to be involved in the central nervous system or meninges and confirmed by MRI or CT, or to have other active central nervous system diseases;
* Patients with plasma cell leukemia or Waldenstrom macroglobulinemia or POEMS syndrome (polyneuropathy, organ enlargement, endocrine disorder, monoclonal protein, and cutaneous disease) or amyloidosis at the time of screening;
* Heart disease: Existing heart failure (NYHA classification ≥II, Appendix 2), unstable angina pectoris, or severe heart disease as determined by the investigator; Myocardial infarction had occurred no more than 6 months before single arthroplasty. Had an episode of unstable angina pectoris, severe arrhythmia as determined by the researchers, or had undergone coronary artery bypass grafting (CABG) no more than 3 months before the single harvest;
* Poor control of hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg) or with hypertensive crisis or hypertensive encephalopathy;
* Patients who had undergone major surgery or plasma separation other than diagnosis or biopsy within 4 weeks prior to the study alone, or who were expected to undergo major surgery during the study period; Note: Patients who plan to undergo surgery under local anesthesia may participate in the study. Kyphoplasty or vertebra osteoplasty are not considered major surgery;
* Receiving thrombolytic, anticoagulant or antiplatelet therapy;
* Infections require intravenous antibiotics or hospitalization;
* Patients with active hepatitis B; Hepatitis C virus (HCV) antibody positive; HIV-positive persons; Syphilis primary screening antibody positive; A) Inactive/asymptomatic patients with carryable, chronic, or active HBV who meet the following criteria are eligible for inclusion: HBV DNA <500 IU/mL (or 2500 copies /mL) at the time of screening.
* Women who are pregnant or lactating;
* The investigator considers that the subject is unsuitable to participate in this clinical study due to any abnormal clinical or laboratory examination or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of all adverse events and serious adverse events | Day 1 through Month 24
  The safety and tolerability of CART-BCMA were evaluated according to the the incidence of all adverse events and serious adverse events
BCMA-CART Maximum Tolerable Dose (MTD) and/or Recommends Dose (RD) | Day 1 through Month 24
  BCMA-CART Maximum Tolerable Dose (MTD) and/or Recommends Dose (RD)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hematology Department of the First Affiliated Hospital of Zhejiang University, Hangzhou
  - Hematology Department of Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided